CLINICAL TRIAL: NCT00176761
Title: A Phase II Trial Assessing Autologous, Tumor-Pulsed Dendritic Cells as a Tumor Vaccine Administered With IL-2 in Patients With Metastatic Colorectal Cancer
Brief Title: Tumor-Pulsed Dendritic Cells Used as a Tumor Vaccine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: University of Michigan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9947; GCRC Protocol #1673
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 (IL-2)

SUMMARY:
This study is being conducted to determine the efficacy, side effects, and toxicity of an investigational vaccine that consists of tumor-pulsed dendritic cells administered with an immune stimulating drug called interleukin-2 (IL-2). Dendritic cells are immune cells that are obtained from a subject's blood and are important in the body's immune response to foreign substances. This study will examine the response of a subject's immune system after receiving several vaccinations containing their own dendritic cells which have been exposed to dead fragments of their cancer cells in the laboratory. This may result in sensitizing a subject's dendritic cells to their cancer cells so that their dendritic cells will react with other cells of the immune system and attack the cancer. It has been shown in the laboratory that dendritic cells exposed to cancer cell fragments can provide lymphocytes (a type of white blood cell) with signals they require in order to become fully activated and acquire the ability to kill cancer cells.

DETAILED DESCRIPTION:
Pretreatment screening: If a subject decides to participate in this study they will first be presented the informed consent document to read and review with the Principal Investigator (or his designee) to go over each aspect of the study and answer any questions. Once the patient has consented, they will first be screened to make sure they meet the eligibility criteria. The screening process is done to make sure that it is appropriate for the subject to participate in this study. This process will include a review of their medical history, a complete physical examination, standard blood tests, an EKG (an electrocardiogram), a chest x-ray and if it is possible for them to become pregnant, a pregnancy test. These tests are normally performed on patients prior to receiving chemotherapy for cancer. In addition to these tests which are normally performed, blood will be obtained for tests which are specific for this investigational study.

These study specific tests include a blood test to determine whether a subject may be infected with the hepatitis B virus or the AIDS virus, and blood tests to determine the ability of their immune system to respond to normal stimulation. A doctor will also order CT scans or nuclear medicine scans to measure the extent of the subject's cancer because the study therapy has a possibility of shrinking the tumor and this will be determined by measuring each subject's disease before and after therapy.

At the time of this initial evaluation subjects will have skin tests that will determine their ability to mount an immune response to infectious agents (such as tetanus, measles, mumps) that they have been exposed to or vaccinated against. If a subject fails to demonstrate a response to all the skin tests, they will not be allowed to participate in this study because such lack of response indicates that their immune system may not respond to the therapy planned in this study.

Vaccine therapy: In order to make a vaccine from a subject's tumor they must have surgical removal of some tumor in order to provide tumor cells. The doctor will determine if a subject has colorectal cancer cells that are easily obtainable. However, if a subject already has an available frozen tumor specimen at the University of Michigan, that may be used for the vaccine preparation instead of undergoing another surgical procedure. This surgery may be done solely for the purpose of participating in this research and may not otherwise benefit a subject. A separate consent form will be required for any surgery a subject undergoes.

The cancer cells obtained from each subject will be taken to the laboratory where they will be separated into single cells, disrupted to make cell fragments, radiated to kill the cells and then mixed with your dendritic cells. The dendritic cells will be obtained from the peripheral blood. Subjects will undergo a procedure called leukapheresis that involves placing a large needle (central line) in a vein in each of their arms. These central lines will be inserted under local anesthesia (subjects will remain awake…only the site of the insertion will be "frozen"). Blood exits from one needle and is processed through a machine that selectively removes one kind of white blood cell and then returns the other elements of the blood back to their body. The leukapheresis procedure generally lasts three to four hours. Following the procedure, the dendritic cells will be cultured in the laboratory to increase the number of dendritic cells. This procedure takes about 2 days.

The tumor-exposed dendritic cell vaccine will be administered as an intradermal (into the skin) injection into a subject's thigh or arm on days 1, 15 and 29 of study treatment. Additionally, they will receive IL-2 by subcutaneous injection daily for 4 days after each vaccination.

Four weeks after their last vaccination, subjects will undergo skin testing to determine if they are reactive to their tumor cells. White blood cells will also be obtained by a second leukapheresis procedure to determine, via research tests in the laboratory, if their circulating immune cells have developed the capacity to respond to their cancer cells. This skin testing and leukapheresis are for research purposes.

Also, 4 weeks after subjects receive their last vaccination, they will have x-rays and/or CT scans done to determine whether their disease has responded to the immune therapy. If their cancer has not worsened or if it has shrunk, then they will be offered the option to receive additional vaccinations using the tumor-pulsed dendritic cells providing that they did not experience severe toxicity with the first series of vaccinations and provided there is enough vaccine material available. The additional vaccinations would be done using the same procedure and schedule as the previous vaccinations until there is evidence that the subject's disease has started to grow or worsen. This includes leukapheresis, vaccination, and IL-2 administration. Re-treatments will be offered until a subject's disease gets worse or tumor cells are no longer available to produce vaccines. A subject's study participation will end with the leukopheresis and tumor evaluation 4 weeks following their last series of vaccinations.

Blood Drawing: The maximum amount of blood, for standard tests and research purposes that will be drawn during the 10 weeks will be a total of 100ccs, which is approximately 20 teaspoons, which is equivalent to approximately 7 tablespoons over the 12 week time period.

The length of time a subject would be on this study is a minimum of nine weeks. If the physician determines that a subject is benefiting from this study, they may continue repeat vaccinations for as long as they continue to have clinical benefit from the study and vaccine is available. During the study, if other therapy alternatives become clinically indicated, they will be discussed with the subject. Also, if there are any significant new findings developed over the course of this research which may affect a subject's willingness to participate, they will be told of them.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have metastatic colorectal cancer. Patients are eligible whether they are previously untreated or had received prior treatment.
2. Patients must have a source of autologous tumor that can be easily harvested. This includes patients with subcutaneous or cutaneous metastases, patients with easily excisable lymph nodes containing metastatic tumor, and patients with malignant pleural effusions or ascites. In addition, some patients who undergo a planned curative operation are found at that time of surgery to be unresectable and these patients could have a sample of tumor resected at that time to be eligible for this study.
3. Karnofsky performance status equal to or greater than 70%.
4. Life expectancy of at least three months.
5. Patients must have evaluable or measurable disease in addition to the disease that will be surgically removed for the purposes of formulating the autologous vaccine.
6. Adequate baseline hematopoietic function:

   1. platelet count equal to or greater than 100,000/mm3
   2. total white blood count equal to or greater than 3,000/mm3
7. Patients must not have received any antineoplastic chemotherapy or immunotherapy for the four weeks preceding entry onto the study (six weeks for nitrosoureas and mitomycin-C).
8. Patients must not have received irradiation for the four weeks prior to entry onto the study.
9. Ability to give informed consent.

Exclusion Criteria

1. Patients may not have received prior antitumor vaccines.
2. History of any autoimmune diseases (e.g. SLE, rheumatoid arthritis, myasthenia gravis).
3. Active infection (bacterial, fungal, or viral), or active bleeding (e.g. hemoptysis, GI bleeding).
4. Pregnancy or lactation; women of childbearing potential and men must use effective contraception during the course of this clinical trial.
5. Uncontrolled angina, arrhythmias, bronchospasm, hypertension, hyperglycemia or hypercalcemia.
6. History of corticosteroid use in the four weeks preceding entry onto the clinical study.
7. Patients who require corticosteroids.
8. Evidence of HIV infection or AIDS and/or testing positive for HBSAg.
9. Any medical or psychiatric illness which in the opinion of the clinical investigators would compromise the patients ability to tolerate this treatment.
10. Patients who require anticoagulation.
11. There is no exclusion for sex or ethnic background.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2000-03; Study Completion 2006-05

PRIMARY OUTCOMES:
To assess the antitumor response of this immunotherapy regimen.

SECONDARY OUTCOMES:
To characterize the immune response (as defined in Section VII) to the tumor-pulsed dendritic cell vaccine combined with IL-2 administration in patients with metastatic colorectal cancer.
To evaluate the toxicity of this treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States